CLINICAL TRIAL: NCT03271827
Title: Apnoeic Oxygenation by Nasal Cannula During Airway Management in Children Undergoing General Anaesthesia: A Pilot Randomised Controlled Trial"
Brief Title: Apnoeic Oxygenation by Nasal Cannula During Airway Management in Children Undergoing General Anaesthesia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: King Abdullah International Medical Research Center (Other); Cardiff University (Other)
Responsible Party: Principal Investigator, Lafi Olayan, Research fellow, University of Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SP15/134
Record Dates: First submitted 2017-08-30; First posted 2017-09-05 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Apnoeic Oxygenation
Keywords: Apnoeic oxygenation; Airway management; Oxygen insufflation; Paediatric general anaesthesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apnoeic oxygenation group (Experimental): Standard airway management + 3 L/min of oxygen by nasal cannula
  Interventions: Device: Apnoeic oxygenation
- Standard care group (No Intervention): Standard airway management

INTERVENTIONS:
Device: Apnoeic oxygenation — 3 L/min of oxygen by nasal cannula during as apnoeic oxygenation during airway management.
  Arms: Apnoeic oxygenation group

SUMMARY:
Airway management is a core clinical skill in anaesthesia. Pre-oxygenation prior to induction of anaesthesia is standard practice to prevent desaturation. Apnoeic oxygenation in adults is effective and prolongs the time to desaturation. The effectiveness of apnoeic oxygenation in the adult is well document, however evidence in the paediatric is lacking. Therefore, the aim of this study was to investigate the effectiveness of apnoeic oxygenation during airway management in children.

This was a pilot randomised controlled trial. Patients were randomised to either receive apnoeic oxygenation or standard care during the induction of anaesthesia. The primary outcome was the duration of safe apnoea, defined as a composite of the time to first event, either time for SpO2 to drop to 92% or time to successfully secure the airway, and the lowest SpO2 observed during airway management. Secondary outcomes were number of patients whose SpO2 dropped below 95% and number of patients whose SpO2 dropped below 92%.

ELIGIBILITY:
Inclusion Criteria:

* Patients were included who were scheduled for elective surgery under general anaesthesia.
* Age: one eight years old.
* ASA I and II only.
* Patients with normal cardiorespiratory function.

Exclusion Criteria:

* Children undergoing dental surgeries in which nasal intubation is needed.
* Patients who suffered from quick drops in oxygen saturation more rapidly than healthy children due to different reasons such as: respiratory and pulmonary diseases, active or recent upper respiratory tract infection, syndromes with cardiopulmonary pathologies, cardiac anomalies, anaemia, depressed respiratory effort, ventilation/perfusion imbalance, Obstructive Sleep Apnoea (OSA), and airway obstruction.
* Patients reported with nasal obstruction.
* Patients with grades of laryngoscopic view (Cormack Lahane) greater than II, which indicates upper airway obstruction.

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Time to first event | Estimated: 10 seconds to 3 minutes
  Time to first event: either time for SpO2 to fall to 92% or time to successfully secure the airway as usual practice without allowing desaturation
The lowest SpO2 observed during airway management | Estimated: 10 seconds to 3 minutes
  The lowest SpO2 observed during airway management

SECONDARY OUTCOMES:
Number of patients whose SpO2 dropped below 95% | Estimated: 10 seconds to 3 minutes
  Number of patients whose SpO2 dropped below 95%
Number of patients whose SpO2 dropped below 92% | Estimated: 10 seconds to 3 minutes
  Number of patients whose SpO2 dropped below 92%

CONTACTS AND LOCATIONS:
Overall Officials: Lafi Olayan, MSc, Principal Investigator — King Abdullah International Research Center (KAIMRC)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weingart SD, Levitan RM. Preoxygenation and prevention of desaturation during emergency airway management. Ann Emerg Med. 2012 Mar;59(3):165-75.e1. doi: 10.1016/j.annemergmed.2011.10.002. Epub 2011 Nov 3. PMID 22050948
- [Background] Baraka AS, Taha SK, Siddik-Sayyid SM, Kanazi GE, El-Khatib MF, Dagher CM, Chehade JM, Abdallah FW, Hajj RE. Supplementation of pre-oxygenation in morbidly obese patients using nasopharyngeal oxygen insufflation. Anaesthesia. 2007 Aug;62(8):769-73. doi: 10.1111/j.1365-2044.2007.05104.x. PMID 17635423
- [Background] Ramachandran SK, Cosnowski A, Shanks A, Turner CR. Apneic oxygenation during prolonged laryngoscopy in obese patients: a randomized, controlled trial of nasal oxygen administration. J Clin Anesth. 2010 May;22(3):164-8. doi: 10.1016/j.jclinane.2009.05.006. PMID 20400000
- [Background] Wimalasena Y, Burns B, Reid C, Ware S, Habig K. Apneic oxygenation was associated with decreased desaturation rates during rapid sequence intubation by an Australian helicopter emergency medicine service. Ann Emerg Med. 2015 Apr;65(4):371-6. doi: 10.1016/j.annemergmed.2014.11.014. Epub 2014 Dec 20. PMID 25536868
- [Background] Taha SK, Siddik-Sayyid SM, El-Khatib MF, Dagher CM, Hakki MA, Baraka AS. Nasopharyngeal oxygen insufflation following pre-oxygenation using the four deep breath technique. Anaesthesia. 2006 May;61(5):427-30. doi: 10.1111/j.1365-2044.2006.04610.x. PMID 16674614
- [Background] Hardman JG, Wills JS, Aitkenhead AR. Factors determining the onset and course of hypoxemia during apnea: an investigation using physiological modelling. Anesth Analg. 2000 Mar;90(3):619-24. doi: 10.1097/00000539-200003000-00022. PMID 10702447
- [Background] Hardman JG, Wills JS. The development of hypoxaemia during apnoea in children: a computational modelling investigation. Br J Anaesth. 2006 Oct;97(4):564-70. doi: 10.1093/bja/ael178. Epub 2006 Jul 27. PMID 16873387
- [Derived] Olayan L, Alatassi A, Patel J, Milton S. Apnoeic oxygenation by nasal cannula during airway management in children undergoing general anaesthesia: a pilot randomised controlled trial. Perioper Med (Lond). 2018 Feb 21;7:3. doi: 10.1186/s13741-018-0083-x. eCollection 2018. PMID 29484172